CLINICAL TRIAL: NCT05974111
Title: COAgulation Disorders in Ischaemic and Haemorrhagic Stroke
Acronym: COADIHS
Status: Recruiting | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Synapse bv (Industry)
Responsible Party: Sponsor
Other Study IDs: Z-2022142
Record Dates: First submitted 2023-05-30; First posted 2023-08-03 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Stroke; Haemorrhagic Stroke; Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Subarachnoid Hemorrhage | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples stored in biobank for full coagulation testing. Moreover cell free DNA methylation will be assessed as marker of neuronal ischemia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Ischemic Stroke: Patients presenting at emergency department / Intensive Care unit with ischemic stroke
  * registration of baseline clinical data
  * registration of baseline blood parameters (in context of standard of clinical care)
  * additional blood sampling at 5 time points during 1st week with the purpose of full coagulation testing and cell free DNA methylation
  Interventions: Diagnostic Test: blood sampling
- Haemorrhagic stroke: Patients presenting at emergency department / Intensive Care unit with haemorraghic stroke (spontaneous intracranial bleeding, no trauma)
  * registration of baseline clinical data
  * registration of baseline blood parameters (in context of standard of clinical care)
  * additional blood sampling at 5 time points during 1st week with the purpose of full coagulation testing and cell free DNA methylation
  Interventions: Diagnostic Test: blood sampling
- Aneursmal Subarachnoid Haemorrhage: Patients presenting at emergency department / Intensive Care unit with aneurysmal subarachnoid haemorrhage
  * registration of baseline clinical data
  * registration of baseline blood parameters (in context of standard of clinical care)
  * additional blood sampling at 5 time points during 1st week with the purpose of full coagulation testing and cell free DNA methylation
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — At 5 time points (D0 (T0),morning after (T0B),D3 (T1),D5 (T2),D7(T3)) blood samples will be drawn next to blood sampling in context of standard of clinical care. A full coagulation and inflammation profile will be obtained as well as cell free DNA methylation

SUMMARY:
In this study the investigators will assess both procoagulant and anticoagulant pathways using thrombin generation and platelet function tests; as well as neuronal ischemia using cell free DNA in all patients presenting with ischaemic and haemorrhagic stroke (including aneurysmal subarachnoid haemorraghe). Also the cross-talk between inflammation and thrombosis, so-called thrombo-inflammation is further investigated. As such the investigators aim to characterise the patient's coagulation profile before administration of any treatment. By assessing these pathways the investigators strive to detect specific markers to predict vital and functional outcome at 3 months in these patients. Finally the investigators may provide new pathophysiological insights in the course of disease following these events that can possibly improve future therapeutic strategies.

DETAILED DESCRIPTION:
In the COADIHS trial the main objective is to map the coagulation profile, both procoagulant and anticoagulant pathways, in patients presenting with acute ischaemic or haemorrhagic stroke.

By assessing these different pathways the investigators aim to detect possible biomarkers of coagulation with predictive value for functional and vital outcome at 3 months.

In different subgroup analyses the investigators try to answer additional research questions as posed by the specific pathophysiology.

Primary Objective:

Mapping the coagulation profile of both procoagulant and anticoagulant pathways together with markers of inflammation and ischemia in patients presenting with all types of acute ischaemic or haemorrhagic stroke, at presentation and during first 7 days of clinical course in order to detect biochemical markers with predictive value of vital and functional outcome at 3 months.

Secondary Objective:

* Detection of culprit underlying thrombophilia in cryptogenic stroke and evaluation of their effect on clinical course and outcome (recurrent stroke).
* Evaluating the interaction between the coagulation profile and pre-stroke medication that works on coagulation pathways.
* To investigate the role of platelets and platelet activation in different pathophysiological mechanisms described in development of delayed cerebral ischemia following aneurysmal subarachnoid haemorrhage (aSAH)(microvessel constriction, thromboinflammation, large artery vasospasm, cortical spreading depolarization)
* To evaluate the role of haemostatic derangements following aSAH as biomarker to predict delayed cerebral ischemia.

ELIGIBILITY:
Inclusion Criteria:

Presenting at the hospital with ischaemic stroke, haemorrhagic stroke, aneurysmal subarachnoid haemorrhage or any other type of non-traumatic, intracranial bleeding

In patients with minor ischemic stroke (NIHSS <= 4) only baseline lab sampling will be performed (T0 and T0B).

Exclusion Criteria:

* Refusal of participation by patient or legal representative
* Traumatic intracranial (subdural, subarachnoid, epidural haematoma) bleeding
* Patients receiving treatment with interference on coagulation (pro / anti) before first sampling: in this group of patients the coagulation assessment at presentation will be excluded, further lab sampling is performed according to protocol.
* Patients categorized as having stroke mimic will be excluded from analysis afterwards

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients presenting at the hospital with ischaemic stroke, haemorrhagic stroke or aneurysmal subarachnoid haemorrhage.
  As our hospital is a referral centre, both referred patients and patients presenting at our emergency department will be screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Functional Outcome Modified rankin scale | 3 months
  Modified Rankin Scale as defined by:
  score 0: no symptoms score 1: No significant disability despite symptoms; able to carry out all usual duties and activities Score 2:Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance Score 3: Moderate disability; requiring some help, but able to walk without assistance Score 4:Moderately severe disability; unable to walk and attend to bodily needs without assistance Score 5: Severe disability; bedridden, incontinent and requiring constant nursing care and attention Score 6:Dead
  With Score 3-6 defined as poor outcome and score 0-2 defined as good outcome
Functional Outcome recurrent stroke | 3 months
  Recurrent stroke during first 3 months
Vital Outcome - all cause mortality | 3 months
  Mortality rate in the participants of all cause at 3 months
Functional Outcome EuroQol-5D | 3 months
  EuroQol-5D questionnaire scoring different aspects of functionality
  In each dimension a scale of 1-5 will be recorded, defined as:
  * mobility
    1. No problems
    2. Slight problems
    3. Moderate problems
    4. Severe problems
    5. 'unable to'
  * self-care
    1. No problems
    2. Slight problems
    3. Moderate problems
    4. Severe problems
    5. 'unable to'
  * usual activities
    1. No problems
    2. Slight problems
    3. Moderate problems
    4. Severe problems
    5. 'unable to'
  * pain/discomfort
    1. No problems
    2. Slight problems
    3. Moderate problems
    4. Severe problems
    5. extreme
  * anxiety / depression
    1. No problems
    2. Slight problems
    3. Moderate problems
    4. Severe problems
    5. extremely
  a global health score will be assessed

SECONDARY OUTCOMES:
ICU Length of stay | 3 months
  duration (days)
Hospital Length of stay | 3 months
  duration (days)
Need for mechanical ventilation in ICU | 3 months
  Yes/No and duration (days)
Need for renal replacement therapy in ICU | 3 months
  YES / NO and duration (days)
Deep vein thrombosis | 3 months
  Yes/No
Need for ventriculo-external drain / ventriculo-peritoneal drain | 3 months
  Yes / No
Rate of delayed cerebral ischemia participants with aneurysmal subarachnoid haemorrhage | 3 months
  Rate of delayed cerebral ischemia in participants with aneurysmal subarachnoid haemorrhage
  * vasospasm: clinical / radiological (transcranial doppler, CT perfusion, MRI)
  * Delayed cerebral ischemia as diagnosed with MRI
Need for decompressive craniectomy | 3 months
  Yes / no
Haemorrhagic transformation of infarction | 3 months
  yes / No
Rebleeding aneurysm in aneurysmal subarachnoid haemorrhage | 3 months
  yes /no
Rate of epilepsy | 3 months
  Both convulsive epileptic episode as non-convulsive epileptic episode. Both clinical diagnosis and elektro-encephalogram
Rate of infection in participants | 3 months
  CNS infection, Pulmonary infection, genito-urinary infection, catheter related blood stream infection,gastro-intestinal infection, skin infection, other infection, bacteriemia, fungaemia
Rate of Intensive Care Aquired weakness (ICUAW) | 3 months
  critical illness myopathy, critical illness polyneuropathy or icu-AW
Rate of diabetes insipidus during first week | 7days
  Diabetes insipidus
Rate of cardiovascular compromise during first week | 7 days
  As defined by use of vasopressors and inotropes / acute heart failure / acute myocardial infarction / cardiac arrest / new arrythmia / use of VA-ECMO
Rate of acute respiratory failure during first week | 7 days
  acute respiratory failure (intubation + mechanical ventilation / non-invasive ventilation / ARDS), need for VV-ECMO / neurogenic pulmonary edema
Rate of Acute kidney injury during first week | 7 days
  acute kidney injury (KDIGO classification)
Rate of enteral feeding (oral/nasograstic) or Total parenteral nutrition during first week | 7 days
  TPN / enteral feeding (oral/nastrogastric)
Rate of Acute liver failure during first week | 7 days
  Acute liver failure
  * INR > 1.5
  * Any grade of hepatic encefalopathy
  * No prior evidence of liver disease
Rate of infection during first week | 7 days
  CNS infection / pulmonary infection / endocarditis / UTI / GI infection /skin infection / blood stream infection
Rate of antiplatelet / anticoagulant therapy during first week | 7 days
  Rate of antiplatelet therapy or anticoagulant therapy in participants

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Stragier, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No